CLINICAL TRIAL: NCT06858098
Title: Outcomes of a Pre-operative Exercise Regimen for Patients Undergoing Hand-assisted Liver Donor Nephrectomy and Transplantation
Brief Title: Outcomes of a Pre-operative Exercise Programme for Live Donor and Recipient Kidney Transplant Patients
Acronym: OPERATe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Gareth Kitchen, Chief Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 316796
Record Dates: First submitted 2025-02-17; First posted 2025-03-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant; Kidney Transplant Donor; Kidney Transplant Recipient
Keywords: live kidney transplant; prehabilitation; wearable devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Entire cohort (Experimental): All participants (both transplant donor and recipients) will be assigned a 6 week graded pre operative outpatient exercise regimen (prehabilitation) delivered by video instruction. Participants will also be monitored 24/7 by a wearable smart device for a total 14 week period (2 week baseline data collection, 6 weeks during prehabilitation and 6 weeks post op).
  Interventions: Other: Exercise programme; Device: Wearable smart device

INTERVENTIONS:
Other: Exercise programme — 6 week pre-operative graded prehabilitation programme, delivered by video and performed by participant up to 4 times a week at home or in a gym setting
Device: Wearable smart device — Participants will wear a wearable smart device (wrist or ring worn) for a period for 14 weeks; 2 weeks prior to prehabilitation, 6 weeks during pre-operative prehabilitation and 6 weeks post operative monitoring,

SUMMARY:
The goal of this clinical trial is to learn if a pre-operative outpatient exercise programme, monitored by a smart wearable device is acceptable to live kidney donor and recipient transplant patients. It will also look at the impact of prehabilitation on post operative outcomes. The main questions it aims to answer are:

Is it feasible for renal transplant patients and live kidney donors to participate in a prehabilitation programme in combination with a piece of wearable technology?

Are transplant outcomes improved by prehabilitation regimens delivered by video instruction?

Are there discernible perioperative digital signatures provided by the wearable that link to surgical outcomes?

Is the quality of perioperative sleep linked to surgical outcomes?

Participants will:

Wear a wrist or ring worn wearable device for a total of 14 weeks (2 week baseline, 6 week pre op and 6 week post op) Engage in a 6 week pre operative exercise programme at home/gym Keep a diary and answer surveys on their experience of the exercise regimen and wearable device

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Live kidney donor or transplant recipient

Exclusion Criteria:

* Deceased donor transplant recipient
* Patient unable to wear or tolerate wearable device
* Unstable angina, recent myocardial infarction, recent cerebrovascular accident or new arrythmia
* Patient declines or is unable to participate in the exercise programme
* Lacks capacity to give informed consent to participate in trial
* Non-English speaking
* No access to a smart device to download application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number days exercise regimen performed and wearable device worn | From enrollment to the end of the study at 14 weeks total
  Acceptability of a prehabiltation programme and wearable device. Is a pre-operative exercise regimen, monitored by a wearable smart device acceptable to live kidney donor and recipient transplant patients? Qualitative data collected through patient surveys and journals. Quantitative measures = number of days exercise performed & number of days wearable device worn

SECONDARY OUTCOMES:
Number of participants with post operative complications | From enrollment to the end of the study at 14 weeks total - complications recorded at 6 week post op follow up
  To assess if prehabilitation programmes have a positive effect on surgical outcomes, quantitative data on the rate and type of post operative complications will be recorded at the standard 6 week post operative patient follow up.
REM Sleep pattern analysis | From enrollment to the end of the study at 14 weeks total when data collection ends
  To assess if there is a link between perioperative sleep patterns and post surgical complications, retrospective analysis of changes in REM vs Non-REM sleep patterns over the 14 week period will be compared to the incidence of post operative complications. REM vs. non-REM data is measured by the wearable device.
Resting heart rate and heart rate variability | From enrollment to the end of the study at 14 weeks total when data collection ends
  Are there discernible perioperative digital signatures (vital signs) recorded by the wearable device that are linked to post-operative outcomes? Retrospective analysis of changes in resting heart rate and heart rate variability, both associated with physiological fitness, will be performed and compared to the incidence of post surgical complications in individual participants (outcome 2)

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Kitchen, Principal Investigator — University of Manchester; Hussein Khambalia, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-11-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT06858098/Prot_000.pdf
  • Informed Consent Form (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT06858098/ICF_001.pdf